CLINICAL TRIAL: NCT00231569
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety and Pharmacodynamics of ISIS 301012 in Hypercholesterolemic Subjects on Stable Statin Therapy
Brief Title: Dose-escalating Safety Study in Subjects on Stable Statin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012CS4; EudraCT No.: 2005-002119-26
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2013-12

CONDITIONS: Hypercholesterolemia
Keywords: LDL-cholesterol; apoB-100; apoB-48
MeSH Terms: conditions — Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort B (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort C (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort D (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort E (Experimental): Loading doses followed by weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort F (Experimental): Loading doses followed by extended weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo
- Cohort G (Experimental): Loading doses followed by extended weekly maintenance doses
  Interventions: Drug: ISIS 301012 or Placebo

INTERVENTIONS:
Drug: ISIS 301012 or Placebo — 30 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, and 29
  Arms: Cohort A
Drug: ISIS 301012 or Placebo — 100 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, and 29
  Arms: Cohort B
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, and 29
  Arms: Cohort C
Drug: ISIS 301012 or Placebo — 300 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, and 29
  Arms: Cohort D
Drug: ISIS 301012 or Placebo — 400 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, and 29
  Arms: Cohort E
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and 85
  Arms: Cohort F
Drug: ISIS 301012 or Placebo — 300 mg subcutaneous injection on days 1, 8, 10, 12, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and 85
  Arms: Cohort G

SUMMARY:
The aim of this study is to assess the safety of varying doses of ISIS 301012 in subjects on Stable statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* On a stable dose of >/= 40 mg Simvastatin or atorvastatin daily for >/= 3 months prior to baseline and expected to remain on this dose for the remainder of the study
* LDL-cholesterol between 2.60 and 5.70 mmol/L (100 and 220 mg/dL), inclusive at screening
* Females not of childbearing potential.

Exclusion Criteria:

* History of CHD or CHD-equivalent (such as diabetes mellitus, or another clinical form of atherosclerotic disease, e.g., peripheral arterial disease, abdominal aortic aneurysm, or symptomatic carotid artery disease)
* Fasting triglyceride >2.26 mmol/L (200 mg/dL) at screening
* Any uncontrolled medical/surgical/psychiatric condition, including conditions that may predispose to secondary hypercholesterolemia
* Current diagnosis or known history of complement deficiency or abnormality
* A positive hepatitis B surface antigen or hepatitis C antibody, or a known positive HIV status
* Current diagnosis or known history of liver disease, or has an ALT >ULN at screening
* Known history of fibromyalgia, myopathy, myositis, rhabdomyolysis, any unexplained muscle pain, or has a CPK >ULN at screening
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin that has been adequately treated
* The advisability of a subject taking any prescription medication (apart from simvastatin or atorvastatin) within 6 weeks prior to screening should be discussed with the Isis Medical Monitor
* Subject unwilling to discontinue taking alternative/herbal medication for the duration of the study
* History of drug abuse within 2 years of screening
* Subject unwilling to limit alcohol consumption for the duration of the study: male subjects to a maximum of 3 drinks (30 g) per day, and <12 drinks (120 g) per week; female subjects to a maximum of 2 drinks (20 g) per day, and <8 drinks (80 g) per week
* Known allergy or hypersensitivity to simvastatin
* Undergoing or has undergone treatment with another investigational drug, biologic agent, or device within 3 months, or 3 half lives, prior to screening, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in LDL-cholesterol from baseline | From baseline measurement

SECONDARY OUTCOMES:
Percent reduction in apoB-100 | From baseline measurement
Percent change in HDL-cholesterol, triglycerides, total cholesterol, non-HDL cholesterol, VLDL plus LDL-cholesterol and LDL-cholesterol particle size and concentration | From baseline measurement
Percent change from baseline in LDL/HDL and apoB-100/apo-A1 ratios | From baseline measurement
AEs, SAEs, physical examination data, vital signs, and laboratory analyzes | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- Auburn, Maine, United States
- Netherlands (4):
  - Amsterdam
  - Leiden
  - Rotterdam
  - Utrecht

REFERENCES:
- [Derived] Akdim F, Stroes ES, Sijbrands EJ, Tribble DL, Trip MD, Jukema JW, Flaim JD, Su J, Yu R, Baker BF, Wedel MK, Kastelein JJ. Efficacy and safety of mipomersen, an antisense inhibitor of apolipoprotein B, in hypercholesterolemic subjects receiving stable statin therapy. J Am Coll Cardiol. 2010 Apr 13;55(15):1611-8. doi: 10.1016/j.jacc.2009.11.069. PMID 20378080